CLINICAL TRIAL: NCT01721759
Title: A Single-Arm Phase 2 Study of Nivolumab (BMS-936558) in Subjects With Advanced or Metastatic Squamous Cell Non-Small Cell Lung Cancer Who Have Received At Least Two Prior Systemic Regimens
Brief Title: Study of Nivolumab (BMS-936558) in Patients With Advanced or Metastatic Squamous Cell Nonsmall-cell Lung Cancer Who Have Received At Least 2 Prior Systemic Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-063; 2012-003965-16 (EudraCT Number)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Squamous Cell Non-small Cell Lung Cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab, 3 mg/kg (Experimental): Participants received nivolumab, 3 mg/kg, intravenously over 60 minutes every 2 weeks (on Day 1 of each cycle) until disease progression, discontinuation due to toxicity, withdrawal of consent, or end of study. Every 2-week treatment period was considered to be a cycle.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
  Other Names: BMS-936558

SUMMARY:
The purpose of the study is to assess the objective response rate (change in tumor size from baseline) in patients with advanced or metastatic squamous cell nonsmall-cell lung cancer treated with Nivolumab (BMS-936558) after failure of 2 prior systemic regimens

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women ≥18 years of age
* Patients with histologically or cytologically documented squamous cell nonsmall-cell lung cancer who present with Stage IIIB/Stage IV disease (according to version 7 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology), or with recurrent or progressive disease following multimodal therapy (radiation therapy, surgical resection, or definitive chemoradiation for locally advanced disease
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Disease progression or recurrence after both a platinum doublet-based chemotherapy regimen and at least 1 additional systemic therapy
* Measurable disease by computed tomography scan/magnetic resonance imaging as per Response Evaluation Criteria in Solid Tumors, volume 1.1

Exclusion Criteria:

* Untreated central nervous system (CNS) metastases. Metastases have been treated and patients neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. In addition, patients must have stopped taking corticosteroids or be taking a stable or decreasing dose of ≤10 mg prednisone daily (or equivalent)
* Carcinomatous meningitis
* Active known or suspected autoimmune disease or interstitial lung disease
* Prior treatment on either arm of study CA209-017 or CA184-104
* Prior therapy with anti-Programmed death-1 (anti-PD-1), anti-Programmed cell death ligand 1 (anti-PD-L1), anti-Programmed cell death ligand 2 (anti-PD-L2), anti-CD137, or anti-Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways
* A condition requiring systemic treatment with corticosteroids or other immunosuppressive medications within 14 days of first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2014-01-22 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (20):
  - University Of California Davis Medical Center, Sacramento, California
  - Va San Diego Healthcare System, San Diego, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute., Atlanta, Georgia
  - Local Institution, Metairie, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Providence Cancer Institute, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Beth Israel Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Providence Oncology And Hematology, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Network Office of Research and Innovation, Allentown, Pennsylvania
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Henry-Joyce Cancer Center, Nashville, Tennessee
  - Oncology Consultants, Pa, Houston, Texas
- France (7):
  - Local Institution, Caen
  - Local Institution, Créteil
  - Local Institution, Pierre-Bénite
  - Local Institution, Rennes
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Cologne
  - Local Institution, München
- Italy (3):
  - Local Institution, Livorno
  - Local Institution, Lucca
  - Local Institution, Terni

REFERENCES:
- [Derived] Dercle L, Fronheiser M, Lu L, Du S, Hayes W, Leung DK, Roy A, Wilkerson J, Guo P, Fojo AT, Schwartz LH, Zhao B. Identification of Non-Small Cell Lung Cancer Sensitive to Systemic Cancer Therapies Using Radiomics. Clin Cancer Res. 2020 May 1;26(9):2151-2162. doi: 10.1158/1078-0432.CCR-19-2942. Epub 2020 Mar 20. PMID 32198149
- [Derived] Rizvi NA, Mazieres J, Planchard D, Stinchcombe TE, Dy GK, Antonia SJ, Horn L, Lena H, Minenza E, Mennecier B, Otterson GA, Campos LT, Gandara DR, Levy BP, Nair SG, Zalcman G, Wolf J, Souquet PJ, Baldini E, Cappuzzo F, Chouaid C, Dowlati A, Sanborn R, Lopez-Chavez A, Grohe C, Huber RM, Harbison CT, Baudelet C, Lestini BJ, Ramalingam SS. Activity and safety of nivolumab, an anti-PD-1 immune checkpoint inhibitor, for patients with advanced, refractory squamous non-small-cell lung cancer (CheckMate 063): a phase 2, single-arm trial. Lancet Oncol. 2015 Mar;16(3):257-65. doi: 10.1016/S1470-2045(15)70054-9. Epub 2015 Feb 20. PMID 25704439
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 117 participants treated.
Period: Treatment Period
Arm/Group | Nivolumab, 3 mg/kg
Started (= Starting Treatment) | 117
Completed (= Continuing in the treatment period) | 0
Not Completed | 117
Not completed — Disease Progression | 85
Not completed — Study drug toxicity | 14
Not completed — Death | 1
Not completed — Adverse event unrelated to study drug | 11
Not completed — Participant request to withdraw | 3
Not completed — Other Reasons | 3
Period: End of Study Period
Arm/Group | Nivolumab, 3 mg/kg
Started | 117
Completed (= continuing in the study) | 0
Not Completed | 117
Not completed — Participant Withdrew Consent | 5
Not completed — Death | 101
Not completed — Lost to Follow-up | 1
Not completed — Other Reasons | 10

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug
Arm/Group | Nivolumab, 3 mg/kg
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (9.11)
Age, Customized [Count of Participants; unit: Participants]
  Younger than 65 years | 58
  At least 65 years and younger than 75 years | 43
  75 years and older | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 69
  Unknown or Not Reported | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 99
  Black or African American | 11
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or other Pacific Islander | 0
  Other | 5
Disease stage [Count of Participants; unit: Participants] — Non-Small Cell Lung Cancer is categorized in 4 Stages (I-IV). I: Cancer located only in lungs and has not spread to any lymph nodes. II: Cancer in the lung and nearby lymph nodes. III: Cancer in the lung and lymph nodes in the middle of the chest. Stage III has two subtypes, IIIA (cancer has spread only to lymph nodes on the same side of the chest where the cancer started) and IIIB (cancer has spread to the lymph nodes on the opposite side of the chest, or above the collar bone). IV: Cancer has spread to both lungs, to fluid in the area around the lungs, or to another part of the body
  Participants
    Stage IIIB | 20
    Stage IV | 97
Cell type [Count of Participants; unit: Participants]
  Squamous cell carcinoma | 117
  Other | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG is a 6-item scale used to assess disease progression, daily functioning, and appropriate treatment and prognosis. Performance status is scored on a scale ranging from 0-5, with (best score) 0=fully active and able to carry on all predisease performance without restriction and (worst score) 5=death.
  Participants
    0 | 26
    1 | 91
    2 | 0
    3 | 0
    4 | 0
Central nervous system metastasis [Count of Participants; unit: Participants]
  Yes | 2
  No | 115

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by Independent Radiology Review Committee (IRC)
Description: ORR is defined as the percentage of participants with best overall response (OR) of confirmed complete response (CR) or partial response (PR) divided by the number of participants who received treatment.
  The IRC-assessed ORR (using RECIST v1.1, to confirm response and based on the IRC global radiology review after incorporation of on-study clinical data) was estimated using a binomial response rate and its corresponding 2-sided 95% exact confidence intervals using the Clopper-Pearson method.
Time Frame: Day 1 of treatment up to approximately 14 months
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nivolumab, 3 mg/kg
Number analyzed (Participants) | 117
Percentage of Participants | 14.5 [8.7 to 22.2]

2. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Investigator
Description: ORR is defined as the percentage of treated participants with confirmed complete response (CR) or partial response (PR) per RECIST 1.1 based on investigator assessment.
  The investigator-assessed ORR is summarized by a binomial response rate and its corresponding two-sided 95% exact CIs using Clopper-Pearson method.
Time Frame: Day 1 of treatment to approximately 101 months
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nivolumab, 3 mg/kg
Number analyzed (Participants) | 117
Percentage of Participants | 15.4 [9.4 to 23.2]

3. Secondary Outcome: Duration of Response (DOR) as Assessed by Investigator
Description: DOR is defined as the time from first confirmed response (CR or PR) per investigator assessment to the date of the first documented tumor progression as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first. Participants who start subsequent therapy without a prior reported progression will be censored at the last evaluable tumor assessments prior to initiation of the subsequent anticancer therapy. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who neither progress nor die will be censored on the date of their last evaluable tumor assessment. Median values of DOR, along with two-sided 95% CI in each treatment group will be computed based on a log-log transformation method.
Time Frame: From the first treatment to the date of the first documented tumor progression or death. Approximately up to 101 months
Population: All treated participants who responded
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab, 3 mg/kg
Number analyzed (Participants) | 18
Months | 16.00 [12.45 to 29.54]

4. Primary Outcome: Duration of Response (DOR) as Assessed by Independent Radiology Review Committee (IRC)
Description: DOR is defined as the time from first confirmed response (CR or PR) per IRC assessment to the date of the first documented tumor progression as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first. Participants who start subsequent therapy without a prior reported progression will be censored at the last evaluable tumor assessments prior to initiation of the subsequent anticancer therapy. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who neither progress nor die will be censored on the date of their last evaluable tumor assessment. Median values of DOR, along with two-sided 95% CI in each treatment group will be computed based on a log-log transformation method.
Time Frame: From the first treatment to the date of the first documented tumor progression or death. Approximately up to 14 months
Population: All confirmed responders per IRC
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab, 3 mg/kg
Number analyzed (Participants) | 17
Months | 12 [6.7 to 19.3]

5. Post Hoc Outcome: Duration of Response (DOR) as Assessed by Independent Radiology Review Committee (IRC)
Description: as for outcome 4
Time Frame: From the first treatment to the date of the first documented tumor progression or death. Approximately up to 21 months
Population: All confirmed responders per IRC
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab, 3 mg/kg
Number analyzed (Participants) | 17
Months | NA [8.31 to NA] — the median and its 95% upper limit were not reached per the Kaplan-Meier method, as the probability in response was still above 50%

ADVERSE EVENTS:
Time Frame: From the first visit to 100 days after last treatment. Approximately up to 101 months
Description: 101 deaths occurred on or before the last disposition date; 7 deaths occurred after the last disposition date
Arm/Group | Nivolumab, 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 108/117
Serious Adverse Events (participants affected / at risk) | 88/117
Other Adverse Events (participants affected / at risk) | 110/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab, 3 mg/kg (N=117)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Pain (General disorders) | 3
Performance status decreased (General disorders) | 1
Pyrexia (General disorders) | 2
Sudden death (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 10
Pulmonary sepsis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain oedema (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 2
Haemorrhage intracranial (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Peripheral nerve paresis (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Urinary tract disorder (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Superior vena cava syndrome (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab, 3 mg/kg (N=117)
Anaemia (Blood and lymphatic system disorders) | 22
Abdominal pain (Gastrointestinal disorders) | 14
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 31
Diarrhoea (Gastrointestinal disorders) | 24
Dry mouth (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 37
Vomiting (Gastrointestinal disorders) | 24
Asthenia (General disorders) | 24
Chest pain (General disorders) | 8
Fatigue (General disorders) | 62
Mucosal inflammation (General disorders) | 7
Oedema peripheral (General disorders) | 16
Pain (General disorders) | 10
Pyrexia (General disorders) | 24
Bronchitis (Infections and infestations) | 11
Pneumonia (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 7
Fall (Injury, poisoning and procedural complications) | 7
Blood creatinine increased (Investigations) | 10
Weight decreased (Investigations) | 19
Decreased appetite (Metabolism and nutrition disorders) | 46
Dehydration (Metabolism and nutrition disorders) | 10
Hypercalcaemia (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 14
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 11
Neuropathy peripheral (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 40
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 17
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.